CLINICAL TRIAL: NCT06049589
Title: Therapeutic Application of Coconut Oil in Oral Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion Clinica Pardinas (Other)
Collaborators: Universidade da Coruña (Other); University Hospital A Coruña (Other)
Responsible Party: Principal Investigator, Simón Pardiñas López, Principal Investigator, Instituto de Investigacion Biomedica de A Coruna
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: 001-FCP
Record Dates: First submitted 2023-09-01; First posted 2023-09-22 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Periodontal Diseases; Periodontal Inflammation; Periodontal Attachment Loss; Periodontitis
MeSH Terms: conditions — Periodontal Diseases; Periodontal Attachment Loss; Periodontitis | interventions — Coconut Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Coconut oil (Experimental): Participants will perform 10-minute vigorous full-mouth rinses once daily after night (2-minute brushing time) brushing. The amount of coconut oil used will be one teaspoon (5 ml). Each participant will be given a container with volume measurement markings. Patients will be provided with the same toothbrush and toothpaste for their dental hygiene 2 times a day. Participants will be asked not to use products containing xylitol, tea, coffee, systemic antibiotics, or topical fluoride during the study. Any participant who violates these rules will be excluded from the study.
  Reevaluation and sampling will be done after 30 days.
  Interventions: Dietary Supplement: Coconut Oil
- Chlorhexidine (Active Comparator): Participants will vigorously rinse their entire mouth with Chlorhexidine 0.12% daily after morning (2 minute brushing time) and evening brushing. The amount of chlorhexidine used will be one teaspoon (5 ml). Each participant will be given a container with volume measurement markings. Patients will be provided with the same toothbrush and toothpaste for their dental hygiene 2 times a day. Participants will be asked not to use products containing xylitol, tea, coffee, systemic antibiotics, or topical fluoride during the study. Any participant who violates these rules will be excluded from the study.
  Reevaluation and sampling will be done after 30 days.
  Interventions: Drug: Chlorhexidine mouthwash
- Water (Placebo Comparator): Participants will vigorously rinse their entire mouth with water daily after morning (2 minute brushing time) and evening brushing. The amount of water used will be one teaspoon (5 ml). Each participant will be given a container with volume measurement markings. Patients will be provided with the same toothbrush and toothpaste for their dental hygiene 2 times a day. Participants will be asked not to use products containing xylitol, tea, coffee, systemic antibiotics, or topical fluoride during the study. Any participant who violates these rules will be excluded from the study.
  Reevaluation and sampling will be done after 30 days.
  Interventions: Other: Water mouthwash

INTERVENTIONS:
Dietary Supplement: Coconut Oil — Coconut oil rinsing
  Arms: Coconut oil
Drug: Chlorhexidine mouthwash — Chlorhexidine rinsing
  Arms: Chlorhexidine
Other: Water mouthwash — Control with water rinsing
  Arms: Water

SUMMARY:
The scientific literature has verified that coconut oil has properties that open perspectives for its application in order to maintain oral health and, in particular, for the treatment of different oral pathologies.

Thus, the purpose of this project is summarized in the following objectives:

1. Determine in vitro the biocompatibility of coconut oil.
2. Determine in vivo the clinical effect of coconut oil as an adjunct treatment for periodontal disease.

DETAILED DESCRIPTION:
Periodontal disease is one of the most prevalent pathologies in humans. In the latest survey on Oral Health in Spain by the Council of Dentists of Spain, it is determined that between 85-94% of the Spanish population over 35 years of age has some problem related to their gums. Severe periodontal diseases, which can lead to tooth loss, affect 15%-20% of middle-aged adults (35-44 years).

One of the most common products used as an antibacterial agent to treat different oral conditions is chlorhexidine and its derivatives. Chlorhexidine exists commercially in different preparations such as mouthwash, toothpaste and gel, among others. Their main drawbacks are that in the long term they stain the teeth and can cause oral lesions, burning sensation and a deterioration in the sensation of taste.

Likewise, various antibiotics, both local and systemic, are used as an adjuvant in the treatment of certain types of gum diseases. Due to the rapid increase in bacterial resistance due to the extensive use of antibiotics, it is important to evaluate alternative antimicrobial agents that can help reduce the use of antibiotics.

Both the coconut and the plant from which this fruit comes are widely used in traditional medicine. Furthermore, the scientific literature on the biological effect of different presentations of this plant (alcoholic extract of coconut shell, coconut water, coconut oil, etc.) has shown, among others, anti-inflammatory activities, analgesic, antioxidant, antifungal, antimicrobial and even antitumor.

There are several hypotheses that suggest that the benefits of using coconut oil can be attributed to the presence of lauric acid, which has the ability to destroy the lipid membrane of microorganisms such as the herpes virus and Gram positive and Gram negative bacteria. Likewise, the viscosity of the oil could inhibit bacterial adhesion and plaque accumulation.

Recent studies describe that oral rinses with coconut oil provide an inhibition in the accumulation of bacterial plaque and plaque-induced gingivitis and a significant reduction of Streptococcus mutans in saliva, suggesting that coconut oil can have a preventive therapeutic application, with fewer adverse effects and lower cost for the maintenance of oral health and treatment of various oral pathologies such as Gingivitis and Periodontitis.

Therefore, the purpose of this study is to determine the effectiveness of coconut oil as an adjunct treatment for periodontal disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients of legal age (18 years) affected by periodontitis with the ability to read, understand and sign the informed consent after having explained the nature of the study, with a willingness to follow protocol requirements
* Diagnosed with periodontal disease stages II, III and IV and grades B and C
* Minimum of 16 natural teeth

Exclusion Criteria:

* Patients who have been treated with antibiotics in the last 4 weeks and who are currently being treated with antibiotics.
* Patients who regularly use gum or candies with xylitol, coconut or coconut derivatives.
* Patients who have received dental cleaning within the last 6 months.
* Pregnant and breastfeeding patients,
* Patients with allergies to coconut, coconut-derived products and chlorhexidine
* Patients with uncontrolled diabetes, uncontrolled high blood pressure, bleeding disorders, liver or kidney disease, heart disease, active cancer, active infectious diseases (other than periodontitis) and patients with a history of local irradiation therapy in the head/neck area.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Probing depth in mm | At 0 days, 30 days and 60 days
  To evaluate the effect of treatment on probing depth reduction.
Bleeding on probing in percentage | At 0 days, 30 days and 60 days
  To evaluate the effect of treatment on reduction of bleeding on probing
Plaque index in percentage | At 0, 30 and 60 days
  To evaluate the effect of treatment on reduction of plaque accumulation
Volatile compounds in breath in ppm of sulphur compounds | At 0, 30 and 60 days
  To evaluate the effect of treatment on the presence of sulphur compounds present on breath
Type of bacteria present on samples from saliva and crevicular fluid using Illumina SBS (Sequencing by synthesis) | At 0, 30 and 60 days
  To evaluate the effect of treatment on the oral microbiome

SECONDARY OUTCOMES:
Patient perception using Visual Analog Scale | At 0, 30 and 60 days
  To evaluate patient perception on the use of the mouthrinse in a scale from 1 to 10 for each question.
Tooth color change measured with the VITA score | At 0, 30 and 60 days
  To evaluate the change on tooth color before and after using the mouthwash.

CONTACTS AND LOCATIONS:
Overall Officials: Simon Pardinas Lopez, DDS, MS, Principal Investigator — Universidade de A Coruña
Locations (1):
- Clinica Medico Dental Pardiñas, A Coruña, A Coruña, Spain

IPD SHARING:
Plan to Share IPD: No